CLINICAL TRIAL: NCT04471545
Title: The Use of Pectoral Nerve Block Type II in Patients Undergoing Trans-axillary Thoracic Outlet Decompression
Brief Title: PECS II Block in Thoracic Outlet Decompression
Acronym: BLOCKTOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Joep Teijink, Professor, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL72737.100.20
Record Dates: First submitted 2020-07-05; First posted 2020-07-15 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Thoracic Outlet Syndrome
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Intervention Model Description: Randomization will be done through Research manager©. This research program has the possibility to create randomisation logs before the start of the trial.
  A random list of numbers will be generated through Research manager© between 0 and 70. If the number is even, the patient will be allocated to the interventional treatment arm (PECS II block). If the number is uneven, the patient will be allocated to the placebo arm. This list will not be changed during the course of this investigation. Randomisation will be performed by an independent pharmacist from the hospital pharmacy before the start of the trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation will be performed by an independent pharmacist from the hospital pharmacy before the start of the trial. This pharmacist has no other task then creating this list and overseeing the preparation of the syringes used in this trial. Syringes will be prepared with ropivacaine or placebo based on this randomisation list. This syringe will be delivered to the preoperative holding with a label that clearly states BLOCKTOS medication, patient name, date of birth and patient number. This procedure makes sure that the patients, surgeons, anaesthesiologist and any other medical personnel are blinded for the randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Intervention arm: PECS II block with ropivacaine
  Interventions: Procedure: Pectoral nerve block type II
- Control group (Placebo Comparator): Control arm: PECS II block with placebo (saline)
  Interventions: Procedure: Pectoral nerve block type II

INTERVENTIONS:
Procedure: Pectoral nerve block type II — A pectoral nerve block type II will be given to the patient after induction. This is performed ultrasound guided

SUMMARY:
Rationale: Postoperative pain management after transaxillary thoracic outlet decompression surgery (TATOD) is difficult. In a retrospective case-control trial, we found evidence that a PECS II block is able to reduce pain and morphine consumption. This may ultimately lead to less morphine induced side-effects and improved patient satisfaction. However, the risk of bias in retrospective research is high. To determine the effect of PECS II in TATOD, a randomized controlled double blinded trial could offer more valuable scientific evidence. Our hypothesis is that a PECS II block will reduce pain, opioid use and opioid induced side-effects in patients undergoing transaxillary TOD (TATOD).

Objective: The aim of the study is to determine the effect of a PECS II block on postoperative pain and opioid use in patients undergoing TATOD. The secondary objective is to determine the effect of a PECS II block on opioid induced side effects such as postoperative nausea and vomitus and the quality of recovery Study design: Single centre randomized controlled double blinded trial Study population: All patients with Neurogenic Thoracic Outlet Syndrome (NTOS) selected for TATOD by the TOS multidisciplinary workgroup and based on the specifications in 2016 SVS reporting standards.

Intervention: The study group will receive a PECS II block with 40 ml ropivacaine 5 mg/ml. The control group will receive a PECS II block with 40 ml NaCL 0.9%.

Main study parameters/endpoints: Primary outcome parameters are postoperative pain using the Numeric Rated Scale (NRS) score assessed at rest and when moving and postoperative morphine-equivalent consumption. Secondary outcome parameters are postoperative Nausea and Vomitus (PONV) and Quality of Recovery questionnaire (QoR-15).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All patients will undergo ultrasound guided injection, after induction of anaesthesia. The administration of the injection does not invoke any extra physical discom-fort. Possible complications include hematoma and pneumothorax, however, the risk is very low (<1%)[1]. In the intervention group, we expect less pain, a reduced need for pain medica-tion and less postoperative nausea and vomitus. We do not expect an altered postoperative course in the control group. Patients will be asked to fill out a questionnaire. Extra blood sam-ples, site visits, physical examinations or other test will not be done in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NTOS
* Selected for a trans-axillary thoracic outlet decompression (TATOD) by the TOS multidisciplinary workgroup.
* Fit for surgery, defined as ASA (American Society of Anesthesiologists) Classification of I, II or III.
* 18 years of age or older
* Sufficient in speaking and writing the Dutch language
* Normal liver and renal function
* Informed consent

Exclusion Criteria:

* Patients with a history of TOD (Redo-surgery)
* Patients with ATOS or VTOS
* ASA ≥ 4
* Kidney or liver failure with contra-indication for NSAID or paracetamol
* Mental retardation
* Pregnancy
* Patients with chronic strong opioid use (>3 administrations per week or continuous transdermal therapy, longer than the last 3 months)
* Allergy to one or more medications used in the study including, ropivacaine, dexamethasone, propofol, sufentanil, succinylcholine, paracetamol, NSAID, morphine, granisetron
* Patients that have trouble expressing themselves in Dutch. Questionnaires are completed by the patients and checked by the nurses. The questionnaire is in Dutch. If there is a language barrier between the questionnaire, the patient or the health care worker, we believe the validity of the answers is questionable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Change in Pain Numeric Rated Scale | Change pain NRS scale is measured at admission, immediately after surgery and every postoperative day in the morning and in the evening from date of admission until the date of discharge
  Pain is measured using the Numeric Rated Scale (NRS) for pain. This is a psychometric response scale in which patients are asked to rate their pain from 0 to 10 (no pain to extreme pain). This scale is a validated and generally accepted tool to measure pain.
Morphine Equivalent Dose (MED) | Total morphine equivalent dose is measured from date of admission until the date of discharge
  Opioid use is measured in Morphine Equivalent Dose (MED). This is a generally accepted tool to quantify opioid use in patients. We will focus on the total opioid consumption.

SECONDARY OUTCOMES:
Postoperative nausea and vomitus (PONV) | measured at admission, immediately after surgery and every postoperative day in the morning and in the evening from date of admission until the date of discharge
  Postoperative nausea and/or vomitus (PONV) will be assessed by yes or no answer.
Quality of Recovery Scale - 15 (QoR-15) | measured at admission, immediately after surgery and every postoperative day in the morning and in the evening from date of admission until the date of discharge
  The QoR-15 is a recently developed and validated patient-reported outcome measurement (PROM) of postoperative quality of recovery.
  Fifteen questions assess five domains of patient-reported health status: pain, physical comfort, physical independence, psychological support and emotional state. The 11-point numerical rating scale leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] van den Broek RJC, Goeteyn J, Houterman S, Bouwman RA, Versyck BJB, Teijink JAW. Interpectoral-pectoserratus plane (PECS II) block in patients undergoing trans-axillary thoracic outlet decompression surgery; A prospective double-blind, randomized, placebo-controlled clinical trial. J Clin Anesth. 2022 Nov;82:110939. doi: 10.1016/j.jclinane.2022.110939. Epub 2022 Jul 27. PMID 35907370